CLINICAL TRIAL: NCT00246428
Title: Motivational Interviewing (MI) for ETOH+ Teens in the ER
Brief Title: Motivational Interviewing for Alcohol-Positive Teens in the Emergency Room
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIAAAMON09892-10; R01AA009892 (NIH); NIH Grant AA09892-10
Record Dates: First submitted 2005-10-27; First posted 2005-10-31 (Estimated); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Alcohol Abuse; Alcohol Dependence
Keywords: Motivational Interviewing; Alcohol Abuse; Alcohol Dependence; Emergency Care Setting
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Intervention Model Description: Two group randomized design

ARMS (2):
- Individual Interventional Inteview (Experimental): 45 minute counseling session
  Interventions: Behavioral: Individual Motivational Interview (IMI)
- Individual Motivational Interview + Family Check UP (Experimental): Same counseling session as Individual Motivational Interview plus a one hour videotaped family assessment, consisting of the parents and the adolescents discussion family beliefs regarding alcohol, and marijuana.
  Interventions: Behavioral: Individual Motivational Interview + Family Check-Up

INTERVENTIONS:
Behavioral: Individual Motivational Interview (IMI) — Individual counseling sessions with emphasis in personal responsibility, exploration of motivation for drinking and review of potential negative consequences. will be evaluated 6, 9, and 12 months
  Other Names: IMI
  Arms: Individual Interventional Inteview
Behavioral: Individual Motivational Interview + Family Check-Up — One hour videotaped session of family assessment
  Other Names: FAsTask
  Arms: Individual Motivational Interview + Family Check UP

SUMMARY:
The purpose of this study is to determine whether motivational interviewing is effective in reducing alcohol consumption and alcohol problems among young adults who present to an Emergency Room.

DETAILED DESCRIPTION:
The long term objectives of this program of research are to develop effective interventions for reducing problem drinking and associated problems among adolescents and young adults and to further enhance intervention approaches by identifying effective elements of treatment derived from cognitive behavioral social learning theory. Current approaches to behavior change in this area frequently rely on school-based primary prevention programs that do not address cessation/reduction issues for adolescents who are already drinking, rarely address motivational issues related to use and abuse, and cannot target school dropouts. Recently, two studies have shown Motivational Interviewing (MI) to be effective with alcohol-involved adolescents when compared to a control or no intervention condition, but have shown greater harm-reduction effects than alcohol consumption effects. In addition, mechanisms of MI have not been elucidated. The major purposes of this study re to compare MI to a minimal contrast condition in which personalized feedback is provided, and to determine if additional booster sessions will enhance outcomes. The population is older adolescents who have been treated in an Emergency Department (ED) following an alcohol-related event. Thus, school dropouts, a high-risk population, will be included in the study. A 2 (MI versus Feedback Only) x 2 (two booster sessions versus no boosters) factorial design will be used to examine whether a MI combined with booster can effectively change subsequent alcohol use and alcohol problems. Experimental manipulations will be evaluated 6, 9, and 12 months after baseline intervention. The study design has several strengths: (1) it will enable an investigation of the main effects of MI versus Feedback Only, providing a more stringent test of the active ingredients of MI than our current competitive segment permitted; (2) it enables an evaluation of the effects of continued contact as a separate factor; and (3) it allows a test of the interaction between baseline intervention type and booster contact. A secondary purpose of the study is to use explicit mediational analyses, tested within a Structural Equation Modeling framework, to examine the hypothesis that stage of change, use of behavioral alcohol reduction strategies, and alcohol treatment seeking will mediate the relationship between intervention and outcome. Finally, the study will determine whether the diagnosis of alcohol abuse or dependence affects responsivity to our intervention. In addition to its potential contribut8ion to theory, the importance of this work is its potential for providing a cos-effective brief intervention at a "teachable moment" to increase high-risk patients' interest in reducing harmful drinking and related risk-taking behaviors.

ELIGIBILITY:
Inclusion Criteria:

1. Admitted to ER
2. Between 18-24 years old
3. Had a blood alcohol concentration (BAC) greater than .01% according to a biochemical test OR self-reported drinking alcohol in the 6 hours prior to the event that caused their hospital visit OR scored 8 or higher on the Alcohol Use Disorders Identification Test (AUDIT)

Exclusion Criteria:

1. Not English-speaking
2. Had a self-inflicted injury
3. In police custody
4. Did not pass a mental status exam

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 125 (Actual)
Dates: Start 2003-01-01 (Actual); Primary Completion 2008-01-31 (Actual); Study Completion 2008-04-30 (Actual)

PRIMARY OUTCOMES:
Alcohol Consumption | 6, 9, and 12 months

SECONDARY OUTCOMES:
Alcohol-related problems (e.g., drinking and driving) | 6, 9, and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Peter Monti, PhD, Principal Investigator — Brown University
Locations (2):
- United States (2):
  - Rhode Island Hospital, Providence, Rhode Island
  - Brown University, Providence, Rhode Island

REFERENCES:
- [Derived] Barnett NP, Apodaca TR, Magill M, Colby SM, Gwaltney C, Rohsenow DJ, Monti PM. Moderators and mediators of two brief interventions for alcohol in the emergency department. Addiction. 2010 Mar;105(3):452-65. doi: 10.1111/j.1360-0443.2009.02814.x. PMID 20402989